CLINICAL TRIAL: NCT02467270
Title: A Randomized, Open-label, Phase 2 Trial of Ponatinib in Patients With Resistant Chronic Phase Chronic Myeloid Leukemia to Characterize the Efficacy and Safety of a Range of Doses
Brief Title: Ponatinib in Participants With Resistant Chronic Phase Chronic Myeloid Leukemia (CP-CML) to Characterize the Efficacy and Safety of a Range of Doses
Acronym: OPTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP24534-14-203; 2014-001617-12 (EudraCT Number); 15/LO/1192 (Registry Identifier: NRES); U1111-1238-0007 (Other Grant/Funding Number: WHO)
Record Dates: First submitted 2015-06-02; First posted 2015-06-10 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Myeloid Leukemia, Chronic, Chronic Phase
Keywords: Chronic Phase Chronic Myeloid Leukemia; Molecular Response; CML; Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms by Histologic Type; Neoplasms; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases; CP-CML
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms by Histologic Type; Neoplasms; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Ponatinib 45 mg (Experimental): Ponatinib 45 mg orally once daily in each 28-day cycle until achievement of ≤1% BCR-ABL1IS up to data cut-off: 31 May 2020. Once ≤1% BCR-ABL1IS was achieved, participants received reduced dose of ponatinib 15 mg orally once daily.
  Interventions: Drug: Ponatinib
- Cohort B: Ponatinib 30 mg (Experimental): Ponatinib 30 mg orally once daily in each 28 day Cycle until achievement of ≤1% BCR-ABL1IS. Once ≤1% BCR-ABL1IS up to data cut-off: 31 May 2020. Once ≤1% BCR-ABL1IS was achieved, participants received reduced dose of ponatinib 15 mg orally once daily.
  Interventions: Drug: Ponatinib
- Cohort C: Ponatinib 15 mg (Experimental): Participants received ponatinib 15 mg orally once daily up to data cut-off: 31 May 2020 in each 28 day Cycle.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Tablet, taken orally once daily.
  Other Names: Iclusig; AP24534

SUMMARY:
The purpose of this study is to characterize the efficacy of ponatinib administered in 3 starting doses (45 mg, 30 mg, and 15 mg daily) in participants with CP-CML who are resistant to prior tyrosine-kinase inhibitor (TKI) therapy or have T315I mutation, as measured by <=1 % Breakpoint Cluster Region-Abelson Transcript Level using International Scale (BCR-ABL1IS) at 12 months.

DETAILED DESCRIPTION:
The drug being tested in this study is ponatinib. This study will characterize the safety and efficacy of ponatinib over a range of 3 starting doses.

The study will enroll 276 participants in 3 cohorts and each cohort will have 92 participants. All the participants will be randomized to receive once-daily oral administration of 1 of 3 starting doses of ponatinib:

* Cohort A: 45 mg ponatinib tablet
* Cohort B: 30 mg ponatinib tablet
* Cohort C: 15 mg ponatinib tablet

The study is designed to consist of 2 periods: 24-cycle Main treatment period and optional treatment continuation period. Participants will be treated with their randomized dose of study drug in the Main Treatment Period until the occurrence of at least one of the following: absence of CHR by 3 months, absence of MCyR at 12 months, absence of <=1% BCR-ABL1IS at 12 months, loss of <=1% BCR-ABL1IS development of intolerance, or completion of all 24 cycles of treatment (whichever occurs first). Following completion of approximately 5 years or following early withdrawal, participants may enter into an optional treatment continuation period.

This multi-center trial will be conducted in the United States, United Kingdom, Republic of Korea, Spain, France, Taiwan, Australia, Canada, Italy, Chile, Japan, Germany, Argentina, Poland, Czech Republic, Denmark, Hong Kong, Portugal, Russia, Singapore, Switzerland, and Sweden. The overall time to participate in this study is approximately 96 months. Participants will make a final visit to the clinic approximately 30 days after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Have chronic phase-chronic myelogenous leukemia/chronic myeloid leukemia (CP-CML) and have received at least two prior tyrosine kinase inhibitor (TKI) therapies and have demonstrated resistance to treatment OR have documented history of presence of T315I mutation after receiving any number of prior TKI.

   o] The diagnosis of chronic myeloid leukemia (CML) will be made using standard hematopathologic and cytogenetic criteria; CP-CML will be defined by all of the following: i <15% blasts in bone marrow ii <30% blasts plus promyelocytes in bone marrow iii <20% basophils in peripheral blood. iv >= 100*10^9/liter (L) platelets (>=100,000/mm^3). v No evidence of extramedullary disease except hepatosplenomegaly vi No prior diagnosis of AP-CML, and BP-CML o] Cytogenetic assessment at screening must demonstrate the BCR-ABL1 fusion by presence of the t(9;22) Philadelphia chromosome.

   i Variant translocations are only allowed provided they meet inclusion criterion 1d.

   o] Resistance to prior TKI therapy is defined as follows (participants must meet at least 1 criterion): i Three months after the initiation of prior TKI therapy: No cytogenetic response (>95% Ph+) or failure to achieve CHR or new mutation ii Six months after the initiation of prior TKI therapy: BCR-ABL1IS >10% and/or Ph+ >65% or new mutation iii Twelve months after the initiation of prior TKI therapy: BCR ABL1IS >10% and/or Ph+ >35% or new mutation iv At any time after the initiation of prior TKI therapy, the development of a new BCR-ABL1 kinase domain mutation(s) v At any time after the initiation of prior TKI therapy, the development of new clonal evolution vi At any time after the initiation of prior TKI therapy, the loss of CHR, or CCyR, or the confirmed loss of MMR in 2 consecutive tests, one of which has a BCR-ABL1IS transcript level of >=1% or new mutation o] >1% of BCR-ABL1IS as shown by real-time polymerase chain reaction
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
3. Have adequate renal function as defined by the following criterion:

   o] Serum creatinine <=1.5*ULN for institution o] Estimated creatinine clearance >=30 milliliter per minute (mL/min) (Cockcroft-Gault formula)
4. Have adequate hepatic function as defined by the following criteria:

   o] Total serum bilirubin <=1.5*ULN, unless due to Gilbert's syndrome o] Alanine transaminase (ALT) <=2.5*ULN, or <=5*ULN if leukemic infiltration of the liver is present o] Aspartate transaminase (AST) <=2.5*ULN, or <=5*ULN if leukemic infiltration of the liver is present
5. Have normal pancreatic status as defined by the following criterion:

   o] Serum lipase and amylase <=1.5*ULN
6. Have normal QT interval corrected (Frederica) (QTcF) interval on screening electrocardiogram (ECG) evaluation, defined as QTcF of <=450 milliseconds (ms) in males or <=470 ms in females.
7. Have a negative pregnancy test documented prior to enrollment (for females of childbearing potential).
8. Agree to use a highly effective form of contraception with sexual partners from randomization through at least 4 months after the end of treatment (for female and male participants who are fertile).
9. Provide written informed consent.
10. Be willing and able to comply with scheduled visits and study procedures.
11. Have recovered from toxicities related to prior anticancer therapy to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 4.0 grade <=1.

Exclusion Criteria:

1. Have used any approved TKIs or investigational agents within 2 weeks or 6 half-lives of the agent, whichever is longer, prior to receiving study drug.
2. Received interferon, cytarabine, or immunotherapy within 14 days, or any other cytotoxic chemotherapy, radiotherapy, or investigational therapy within 28 days prior to receiving the first dose of ponatinib, or have not recovered (>grade 1 by NCI CTCAE, version 4.0) from AEs (except alopecia), due to agents previously administered.
3. Have undergone autologous or allogeneic stem cell transplant <60 days prior to receiving the first dose of ponatinib; have any evidence of ongoing graft-versus-host disease (GVHD) or GVHD requiring immunosuppressive therapy.
4. Are being considered for hematopoietic stem cell transplant (HSCT) within 6-12 months of enrollment (note: ponatinib is not to be used as a bridge to HSCT in this trial).
5. Are taking medications with a known risk of Torsades de Pointes.
6. Have previously been treated with ponatinib.
7. Have active CNS disease as evidenced by cytology or pathology; in the absence of clinical CNS disease, lumbar puncture is not required. History itself of CNS involvement is not exclusionary if CNS has been cleared with a documented negative lumbar puncture.
8. Have clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

   o] Any history of myocardial infarction (MI), unstable angina, cerebrovascular accident, or Transient Ischemic Attack (TIA) o] Any history of peripheral vascular infarction, including visceral infarction o] Any revascularization procedure, including the placement of a stent o] Congestive heart failure (CHF) (New York Heart Association [NYHA] class III or IV) within 6 months prior to enrollment, or left ventricular ejection fraction (LVEF) less than lower limit of normal, per local institutional standards, within 6 months prior to enrollment o] History of clinically significant (as determined by the treating physician) atrial arrhythmia or any history of ventricular arrhythmia o] Venous thromboembolism, including deep venous thrombosis or pulmonary embolism, within 6 months prior to enrollment
9. Have uncontrolled hypertension (that is, >150 and >90 for systolic blood pressure (SBP) and diastolic blood pressure (DBP) respectively). Participants with hypertension should be under treatment at study entry to ensure blood pressure control. Those requiring 3 or more antihypertensive medications should be discussed with the medical monitor.
10. Have poorly controlled diabetes defined as HbA1c values of >7.5%. Participants with preexisting, well-controlled diabetes are not excluded.
11. Have a significant bleeding disorder unrelated to CML.
12. Have a history of alcohol abuse.
13. Have a history of either acute pancreatitis within 1 year of study enrollment or of chronic pancreatitis.
14. Have malabsorption syndrome or other gastrointestinal illness that could affect oral absorption of study drug.
15. Have a history of another malignancy, other than cervical cancer in situ or basal cell or squamous cell carcinoma of the skin; the exception is if participants have been disease-free for at least 5 years, and are deemed by the investigator to be at low risk for recurrence of that malignancy.
16. Are pregnant or lactating.
17. Have undergone major surgery (with the exception of minor surgical procedures, such as catheter placement or BM biopsy) within 14 days prior to first dose of ponatinib.
18. Have an active infection which requires intravenous antibiotics.
19. Have a known history of human immunodeficiency virus infection; testing is not required in the absence of prior documentation or known history.
20. Have any condition or illness that, in the opinion of the investigator, would compromise participant safety or interfere with the evaluation of the drug.
21. Have hypersensitivity to the ponatinib active substance or to any of its inactive ingredients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2025-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Clinical Science, Study Director — Takeda
Locations (86):
- United States (16):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Indiana Blood & Marrow Transplantation, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Michigan Medicine, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center - New York, New York, New York
  - NewYork-Presbyterian Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Taussig Cancer Institute Main Campus, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
- Argentina (3):
  - Fundaleu, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital General de Agudo Jose Maria Ramos Mejia, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano La Plata, La Plata, Buenos Aires
- Australia (2):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Canada (3):
  - Princess Margaret Hospital - Toronto, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Saskatchewan Cancer Agency, Regina, Saskatchewan
- Chile (2):
  - Centro de Investigaciones Clinicas Vina del Mar, Viña del Mar, Región de Valparaíso
  - Hospital del Salvador, Providencia, Santiago Metropolitan
- Czechia (2):
  - Ustav Hematologie a Krevni Transfuze Praha, Prague, Prague
  - Fakultni Nemocnice Olomouc, Olomouc
- Aarhus University Hospital, Aarhus C, \Aarhus, Denmark
- France (8):
  - Centre de Lutte Contre le Cancer - Institut Bergonie, Bordeaux, Aquitaine
  - Centre Hospitalier Regional Universitaire de Lille, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Nancy Hopital de Brabois, Vandœuvre-lès-Nancy, Lorraine
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse, Midi-pyrenees
  - Center Hospitalier Universitaire d'Angers, Angers, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Nantes Hotel Dieu, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Poitou-charentes
  - Centre Hospitalier Universitaire de Nice Hopital l'Archet, Nice, Provence-Alpes-Côte d'Azur Region
- Germany (8):
  - Universitaetsklinikum Heidelberg, Mannheim, Baden-Wurttemberg
  - Universitatsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitatsmedizin Rostock, Rostock, Mecklenburg-Vorpommern
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitatsklinikum Jena, Jena, Thuringia
  - Charite Universitatsmedizin Berlin, Berlin
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
- Queen Mary Hospital, Hong Kong, Hong Kong
- Italy (7):
  - Azienda Ospedaliera San Gerardo di Monza, Monza, Monza E Brianza
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro, Pesaro E Urbino
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele, Catania
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Azienda Sanitaria Locale di Pescara Ospedale Civile Dello Spirito Santo, Pescara
  - Sapienza Universita Di Roma, Roma
  - AOUI - Ospedale Policlinico "Giambattista Rossi" di Borgo Roma, Verona
- Poland (5):
  - Malopolskie Centrum Medyczne, Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz, Łódź Voivodeship
- Portugal (2):
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, Lisbon
  - Centro Hospitalar Sao Joao, Porto
- Russia (9):
  - Rostov State Medical University, Rostov-on-Don, Rostov Oblast
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - GBUZ Moscow Clinical Scientific Center DZM, Moscow
  - Russian Academy of Medical Science, Moscow
  - FGU Russian Scientific Research Institute of Hematology and Transfusiology, Saint Petersburg
  - Almazov Federal North-West Medical Research Centre of Department of Health of Russian Federation, Saint Petersburg
  - Samara State Medical University, Samara
  - Saratov State Medical University, Saratov
- Singapore General Hospital, Singapore, Singapore
- The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, South Korea
- Spain (6):
  - Hospital Regional Universitario Carlos Haya, Málaga, Andalusia
  - Hospital Universitario de Gran Canaria Doctor Nergrin, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Akademiska Sjukhuset, Uppsala, Sweden
- University Hospital Zurich, Zurich, Switzerland
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (6):
  - Royal Liverpool University Hospital NHS Trust, Liverpool, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Imperial College Healthcare NHS Trust, London, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Churchill Hospital, Oxford, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Kantarjian HM, Jabbour E, Deininger M, Abruzzese E, Apperley J, Cortes J, Chuah C, DeAngelo DJ, DiPersio J, Hochhaus A, Lipton J, Nicolini FE, Pinilla-Ibarz J, Rea D, Rosti G, Rousselot P, Shah NP, Talpaz M, Srivastava S, Ren X, Mauro M. Ponatinib after failure of second-generation tyrosine kinase inhibitor in resistant chronic-phase chronic myeloid leukemia. Am J Hematol. 2022 Nov;97(11):1419-1426. doi: 10.1002/ajh.26686. Epub 2022 Aug 30. PMID 36054756
- [Derived] Cortes J, Apperley J, Lomaia E, Moiraghi B, Undurraga Sutton M, Pavlovsky C, Chuah C, Sacha T, Lipton JH, Schiffer CA, McCloskey J, Hochhaus A, Rousselot P, Rosti G, de Lavallade H, Turkina A, Rojas C, Arthur CK, Maness L, Talpaz M, Mauro M, Hall T, Lu V, Srivastava S, Deininger M. Ponatinib dose-ranging study in chronic-phase chronic myeloid leukemia: a randomized, open-label phase 2 clinical trial. Blood. 2021 Nov 25;138(21):2042-2050. doi: 10.1182/blood.2021012082. PMID 34407543
- See also: Iclusig® (ponatinib) US Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2014/203469s009lbl.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 61 investigative sites in the Argentina, Austria, Chile, Denmark, France, United Kingdom, Hong Kong, Italy, Japan, Poland, Russia, Singapore, Korea, Republic of, Spain, Sweden, Taiwan, Province Of China, and United States from 30 June 2015 and up to data cut-off: 31 May 2020. The study is ongoing.
Pre-assignment Details: Participants with diagnosis of chronic phase-chronic myelogenous leukemia (CP-CML) who received at least 2 prior tyrosine kinase inhibitor (TKI) therapies were enrolled in 1:1:1 ratio in 3 cohorts: ponatinib: 45 mg (Cohort A); 30 mg (Cohort B); or 15 mg (Cohort C). Participants who started at 45/30 mg received mandatory dose reduction of their daily dose to 15 mg upon achievement of ≤1% breakpoint cluster region-Abelson 1 transcript level as measured by International Scale (BCR-ABL1IS).
Period: Overall Study
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Started | 94 | 95 | 94
Treated (Safety Population) (Included all participants who received at least one dose of study drug.) | 94 | 94 | 94
Completed | 0 | 0 | 0
Not Completed | 94 | 95 | 94
Not completed — Participants Never Treated | 0 | 1 | 0
Not completed — Ongoing | 50 | 41 | 43
Not completed — Adverse Event | 16 | 15 | 14
Not completed — Progressive Disease | 7 | 7 | 4
Not completed — Death | 2 | 0 | 2
Not completed — Lack of Efficacy | 12 | 18 | 23
Not completed — Non-compliance With Study Drug | 0 | 2 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Physician Decision | 0 | 4 | 1
Not completed — Withdrawal by Subject | 4 | 3 | 5
Not completed — Reason not Specified | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg | Total
Number analyzed (Participants) | 94 | 94 | 94 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (14.77) | 48.5 (12.90) | 48.8 (12.71) | 48.3 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 56 | 41 | 141
  Male | 50 | 38 | 53 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 26 | 20 | 68
  Not Hispanic or Latino | 70 | 67 | 72 | 209
  Unknown or Not Reported | 2 | 1 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 16 | 12 | 15 | 43
  Race: Black or African American | 1 | 2 | 3 | 6
  Race: White | 73 | 77 | 72 | 222
  Race: Unknown | 0 | 1 | 3 | 4
  Race: Other | 2 | 1 | 0 | 3
  Race: Missing | 2 | 1 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 15 | 16 | 7 | 38
  Austria | 0 | 0 | 2 | 2
  Chile | 7 | 9 | 9 | 25
  Denmark | 0 | 0 | 1 | 1
  France | 2 | 1 | 2 | 5
  United Kingdom | 1 | 4 | 7 | 12
  Hong Kong | 1 | 3 | 2 | 6
  Italy | 0 | 3 | 0 | 3
  Japan | 5 | 2 | 4 | 11
  Poland | 4 | 6 | 5 | 15
  Russia | 38 | 31 | 38 | 107
  Singapore | 4 | 3 | 2 | 9
  Korea, Republic Of | 0 | 3 | 2 | 5
  Spain | 2 | 1 | 2 | 5
  Sweden | 1 | 2 | 2 | 5
  Taiwan, Province Of China | 4 | 1 | 2 | 7
  United States | 10 | 9 | 7 | 26
Weight [Mean (Standard Deviation); unit: kg] | 78.14 (20.841) | 77.56 (18.375) | 76.71 (17.434) | 77.47 (18.879)
Height [Mean (Standard Deviation); unit: meter] — Population: Number analyzed is the number of participants with data available for height at Baseline.
  meter
    number analyzed (Participants) | 94 | 91 | 92 | 277
    (all) | 1.68 (0.104) | 1.68 (0.098) | 1.68 (0.090) | 1.68 (0.097)
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Score [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity). Only categories with data are reported.
  Participants
    Score= 0 | 74 | 73 | 72 | 219
    Score= 1 | 19 | 20 | 22 | 61
    Score= 2 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Molecular Response (MR2: <=1% Breakpoint Cluster Region-Abelson Transcript Level) as Measured by the International Scale (BCR-ABL1IS) at Month 12
Description: MR2 is defined as a ratio of reverse transcribed transcript of BCR-ABL to ABL <=1% Breakpoint Cluster Region-Abelson Transcript Level as Measured by the International Scale (BCR-ABL1IS), equivalent to a 2-log reduction in transcript.
Time Frame: 12 months after the first dose of study treatment
Population: ITT Population included all participants who were randomized and for whom BCR-ABL1IS could be measured (ie, participants who had the b2a2/b3a2 transcript type), regardless of whether they received the assigned study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 93 | 93 | 91
percentage of participants | 44.1 [33.8 to 54.8] | 29.0 [20.1 to 39.4] | 23.1 [14.9 to 33.1]

2. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR/MR3)
Description: MMR/MR3 is defined as a ratio of reverse transcribed transcript of BCR-ABL to ABL ≤0.1% on the international scale (equivalent to a 3-log reduction in transcript).
Time Frame: 12 months after the first dose of study treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 93 | 93 | 91
percentage of participants | 17.2 | 20.4 | 16.5

3. Secondary Outcome: Percentage of Participants With Major Cytogenetic Response (MCyR)
Description: MCyR is defined as percentage of participants with complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR). Cytogenetic response is the percentage of Philadelphia chromosome positive (Ph+) metaphases in bone marrow (BM). Response is further defined as MCyR: CCyR or PCyR, where CCyR: 0% Ph + metaphases; PCyR: >0 to 35% Ph + metaphases.
Time Frame: 12 months after the first dose of study treatment
Population: ITT Cytogenetic Population included all participants who were randomized and had a cytogenetic assessment at Baseline with ≥20 metaphases examined, regardless of whether they received the assigned study drug. Overall number analyzed are participants with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 91 | 90 | 89
percentage of participants | 48.4 [37.7 to 59.1] | 27.8 [18.9 to 38.2] | 43.8 [33.3 to 54.7]

4. Secondary Outcome: Duration of Major Molecular Response (MMR/MR3)
Description: Duration of MMR/MR3 is defined as the interval between the first assessment at which the criteria for <=0.1% MMR are met until the earliest date at which loss of <=0.1% MMR occurs, or the criteria for progression are met. Progression to accelerated phase (AP) is defined as: >= 15% and <30% blasts in peripheral blood or bone marrow or >=20% basophils in peripheral blood or bone marrow or >=30% blasts + promyelocytes in peripheral blood or bone marrow (but <30% blasts) or <100*109 platelets per liter (/L) in peripheral blood unrelated to therapy or cytogenetic, genetic evidence of clonal evolution, and no extramedullary disease. Progression to blast Phase (BP) is defined as: >=30% blasts in peripheral blood or bone marrow or extramedullary disease other than hepatosplenomegaly.
Time Frame: Baseline up to approximately 8 years
Reporting Status: Not Posted, anticipated posting 2025-06

5. Secondary Outcome: Percentage of Participants With Adjusted Incidence Rates for Treatment Emergent Arterial Occlusive Events (AOEs), Venous Thrombotic Events (VTEs), Adverse Events (AEs), and Serious AEs (SAEs)
Description: Percentage of participants with adjusted incidence rates who developed AOEs and VTEs were categorized according to arterial occlusive events and venous thrombotic events. AE is any untoward medical occurrence in participant administered medicinal investigational drug. Untoward medical occurrence does not necessarily have to have causal relationship with treatment. SAE is any untoward medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation of present hospitalization; results in persistent or significant disability/incapacity; is congenital anomaly/birth defect/is medically important event that may not be immediately life-threatening/result in death or hospitalization, but may jeopardize participant/may require intervention to prevent one of other outcomes listed in definition above, or involves suspected transmission via a medicinal product of an infectious agent.
Time Frame: From first dose up to 30 days after last dose of the study drug up to data cut-off date: 31 May 2020 (Up to approximately 5 years)
Population: Safety Population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 94 | 94 | 94
percentage of participants
  AOEs | 9.6 | 5.3 | 3.2
  VTEs | 1.1 | 0 | 0
  AEs | 100.0 | 93.6 | 94.7
  SAEs | 34.0 | 25.5 | 33.0

6. Secondary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR)
Description: Cytogenetic response is defined as the percentage of Ph+ metaphases in bone marrow (peripheral blood may not be used), with a review of a minimum of 20 metaphases. CCyR is defined as 0% Ph+ metaphases.
Time Frame: Month 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 91 | 90 | 89
percentage of participants | 34.1 | 17.8 | 29.2

7. Secondary Outcome: Percentage of Participants With Molecular Response 4 (MR4) and Molecular Response (MR4.5)
Description: MR4 is defined as <=0.01% BCR-ABL1IS. MR 4.5 is defined as <=0.0032% BCR-ALB1IS.
Time Frame: Up to approximately 8 years
Reporting Status: Not Posted, anticipated posting 2025-06

8. Secondary Outcome: Percentage of Participants With Molecular Response 1 (MR1)
Description: MR1 is defined as percentage of participants achieving a ratio of <=10% Breakpoint Cluster Region-abelson (BCR-ABL1) transcripts on the international scale. MR1 is molecular response with 1-log reduction in transcript.
Time Frame: 3 months after the first dose of study treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 93 | 93 | 91
percentage of participants | 52.7 | 44.1 | 42.9

9. Secondary Outcome: Percentage of Participants With Complete Hematologic Response (CHR)
Description: CHR is defined as achieving all of the following measurements: white blood cells (WBC) <= institutional upper limit of normal (ULN), platelets <450,000 per cubic millimeter (/mm^3), no blasts or promyelocytes in peripheral blood, <5% myelocytes plus metamyelocytes in peripheral blood, basophils in peripheral blood <5%, and no extramedullary involvement (including no hepatomegaly or splenomegaly).
Time Frame: 3 months after the first dose of study treatment
Population: All randomized participants were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 94 | 95 | 94
percentage of participants | 87.2 [78.8 to 93.2] | 81.1 [71.7 to 88.4] | 81.9 [72.6 to 89.1]

10. Secondary Outcome: Percentage of Participants With Treatment Emergent AEs Leading to Treatment Discontinuation, Dose Reduction and Dose Interruption
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to data cut-off: 31 May 2020 (Approximately 5 years)
Population: Safety Population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 94 | 94 | 94
percentage of participants
  TEAEs Leading to Treatment Discontinuation | 19.1 | 16.0 | 13.8
  TEAEs Leading to Dose Reduction | 45.7 | 35.1 | 31.9
  TEAEs Leading to Dose Interruption | 71.3 | 61.7 | 58.5

11. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response (DOR) of <=1% BCR-ABL1 IS (MR2) at Months 12 and 24
Description: DOR (≤1% BCR-ABL1IS) is defined as interval between first assessment at which criteria for ≤1% BCR-ABL1IS are met until earliest date at which loss of ≤1% BCR-ABL1IS occurs, or criteria for progression accelerated phase (AP) or blast Phase (BP) of chronic myeloid leukemia (CML) are met. Loss of ≤1% BCR-ABL1IS is an increase to >1% of BCR-ABL1IS. Progression to AP: ≥15% and <30% blasts in peripheral blood or bone marrow or ≥20% basophils in peripheral blood or bone marrow or ≥30% blasts + promyelocytes in peripheral blood or bone marrow (but <30% blasts) or <100*109 platelets per liter in peripheral blood unrelated to therapy or cytogenetic, genetic evidence of clonal evolution, and no extramedullary disease. Progression to BP: ≥30% blasts in peripheral blood or bone marrow or extramedullary disease other than hepatosplenomegaly. Kaplan-Meier method was used for analysis of percentage of participants who achieved DOR of 12 and 24 months.
Time Frame: 12 and 24 months after the first dose of study treatment
Population: ITT Population included all participants who were randomized and for whom BCR-ABL1IS could be measured (ie, participants who had the b2a2/b3a2 transcript type), regardless of whether they received the assigned study drug. Data is reported for responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 52 | 35 | 33
percentage of participants
  Month 12 | 79.13 [64.5 to 88.3] | 79.20 [61.2 to 89.5] | 90.10 [72.4 to 96.7]
  Month 24 | 73.17 [57.0 to 84.1] | 75.60 [56.9 to 87.0] | 90.10 [72.4 to 96.7]

12. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response (DOR) of Major Molecular Response (MMR/MR3)
Description: Duration of MMR/MR3 is defined as interval between first assessment at which criteria for MMR are met until earliest date at which loss of MMR occurs, or criteria for progression (progression to AP or BP of CML) are met. Participants remaining in MMR will be censored at last date at which criteria for MMR are met. Loss of MMR is an increase to >0.1% of BCR-ABL1IS. Progression to AP: >= 15% and <30% blasts in peripheral blood or bone marrow or >=20% basophils in peripheral blood or bone marrow or >=30% blasts+promyelocytes in peripheral blood or bone marrow (but <30% blasts) or <100*109 platelets/L in peripheral blood unrelated to therapy or cytogenetic, genetic evidence of clonal evolution, and no extramedullary disease. Progression to BP: >=30% blasts in peripheral blood or bone marrow or extramedullary disease other than hepatosplenomegaly. Kaplan-Meier method was used for analysis of percentage of participants who achieved DOR of 12 and 24 months.
Time Frame: 12 and 24 months after the first dose of study treatment
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 32 | 24 | 21
percentage of participants
  Month 12 | 88.97 [69.5 to 96.3] | 93.33 [61.3 to 99.0] | 94.74 [68.1 to 99.2]
  Month 24 | 88.97 [69.5 to 96.3] | 84.00 [48.7 to 95.9] | 94.74 [68.1 to 99.2]

13. Secondary Outcome: Duration of Response in Responders
Description: Duration of response in "responders" is defined as any participants who achieved ≤1% BCR-ABL1IS at any time during the study. Responders are defined as those participants who meet all of the following: are randomized and treated, respond at 12 months after the initiation of study treatment, and undergo baseline polymerase chain reaction (PCR) assessment.
Time Frame: Baseline up to data cut-off: 31 May 2020 (Approximately 5 years)
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 52 | 35 | 33
months | NA [26.9 to NA] — Median and upper limit of 95% confidence interval (CI) was not estimable as participants were censored. | NA [27.3 to NA] — Median and upper limit of 95% CI was not estimable as participants were censored. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI was not estimable as participants were censored.

14. Secondary Outcome: Time to Response
Description: Time to response was defined as the time interval from the date of the first dose of the study drug until the initial observation of CR or PR for participants with confirmed CR/PR. CR for target lesion: disappearance of all extranodal lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. CR for non-target lesion: Disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis) and norrmalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the Baseline sum diameters.
Time Frame: Baseline up to data cut-off: 31 May 2020 (Approximately 5 years)
Population: ITT Population included all participants who were randomized and for whom BCR-ABL1IS could be measured (ie, participants who had the b2a2/b3a2 transcript type), regardless of whether they received the assigned study drug. Data is reported for the responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 52 | 35 | 33
months | 6.00 [3.1 to 6.0] | 3.04 [3.0 to 6.0] | 6.04 [3.0 to 9.1]

15. Secondary Outcome: Percentage of Participants With Progression to Accelerated Phase (AP)-Chronic Myeloid Leukemia (CML) or Blast Phase (BP)-CML
Description: Progression to AP is defined as: >=15% and <30% blasts in peripheral blood or bone marrow or >=20% basophils in peripheral blood or bone marrow or >=30% blasts + promyelocytes in peripheral blood or bone marrow (but <30% blasts) or <100*109 platelets/L in peripheral blood unrelated to therapy or cytogenetic, genetic evidence of clonal evolution, and no extramedullary disease. Progression to BP is defined as: >=30% blasts in peripheral blood or bone marrow or extramedullary disease other than hepatosplenomegaly.
Time Frame: From first dose date of study treatment up to data cut-off: 31 May 2020 (Approximately 5 years)
Population: All randomized participants were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 94 | 95 | 94
percentage of participants
  Progressed to AP-CML | 10.6 | 9.5 | 11.7
  Progressed to BP-CML | 3.2 | 1.1 | 1.1

16. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the interval between the first dose date of study treatment and the first date at which the criteria for progression are met (progression to the AP or BP of CML), or death due to any cause, censored at the last response assessment. Progression to AP is defined as: >=15% and <30% blasts in peripheral blood or bone marrow or >=20% basophils in peripheral blood or bone marrow or >=30% blasts + promyelocytes in peripheral blood or bone marrow (but <30% blasts) or <100*109 platelets/L in peripheral blood unrelated to therapy or cytogenetic, genetic evidence of clonal evolution, and no extramedullary disease. Progression to BP is defined as: >=30% blasts in peripheral blood or bone marrow or extramedullary disease other than hepatosplenomegaly.
Time Frame: Up to data cut-off: 31 May 2020 (Up to approximately 5 years)
Population: All randomized participants were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 94 | 95 | 94
months | NA [NA to NA] — Median, Lower limit and Upper limit of 95% confidence interval was not estimable due to low number of participants with event. | NA [35.6 to NA] — Median and Upper limit of 95% confidence interval was not estimable due to low number of participants with event. | 45.64 [38.7 to NA] — Upper limit of 95% confidence interval was not estimable due to low number of participants with event.

17. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval between the first does of study treatment and death due to any cause, censored at the last contact date when the participant was alive.
Time Frame: Up to data cut-off: 31 May 2020 (Up to approximately 5 years)
Population: All randomized participants were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
Number analyzed (Participants) | 94 | 95 | 94
months | NA [NA to NA] — Median, Lower limit and Upper limit of 95% confidence interval was not estimable due to low number of participants with event. | NA [NA to NA] — Median, Lower limit and Upper limit of 95% confidence interval was not estimable due to low number of participants with event. | NA [NA to NA] — Median, Lower limit and Upper limit of 95% confidence interval was not estimable due to low number of participants with event.

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after last dose of the study drug up to data cut-off: 31 May 2020 (Up to approximately 5 years)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. All cause-mortality was collected for all randomized participants. Serious and other adverse events was collected for participants from Safety Population who received at least 1 dose of study drug.
Arm/Group | Cohort A: Ponatinib 45 mg | Cohort B: Ponatinib 30 mg | Cohort C: Ponatinib 15 mg
All-Cause Mortality (participants affected / at risk) | 8/94 | 7/95 | 8/94
Serious Adverse Events (participants affected / at risk) | 32/94 | 24/94 | 31/94
Other Adverse Events (participants affected / at risk) | 92/94 | 85/94 | 86/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Ponatinib 45 mg (N=94) | Cohort B: Ponatinib 30 mg (N=94) | Cohort C: Ponatinib 15 mg (N=94)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 3
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Coeliac artery stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 0 | 1
Sudden death (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 2
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0
Age-related macular degeneration (Eye disorders) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Mesenteric vascular Insufficiency (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Ponatinib 45 mg (N=94) | Cohort B: Ponatinib 30 mg (N=94) | Cohort C: Ponatinib 15 mg (N=94)
Thrombocytopenia (Blood and lymphatic system disorders) | 40 | 36 | 35
Neutropenia (Blood and lymphatic system disorders) | 28 | 22 | 23
Anaemia (Blood and lymphatic system disorders) | 20 | 17 | 16
Leukopenia (Blood and lymphatic system disorders) | 5 | 4 | 7
Lipase increased (Investigations) | 19 | 17 | 12
Platelet count decreased (Investigations) | 11 | 9 | 10
Alanine aminotransferase increased (Investigations) | 21 | 6 | 16
Aspartate aminotransferase increased (Investigations) | 13 | 3 | 8
Blood alkaline phosphatase increased (Investigations) | 5 | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 12 | 9 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 7 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 5 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 6 | 3 | 1
Constipation (Gastrointestinal disorders) | 10 | 11 | 14
Abdominal pain (Gastrointestinal disorders) | 9 | 8 | 7
Abdominal pain upper (Gastrointestinal disorders) | 8 | 10 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 20 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 3
Hypertension (Vascular disorders) | 26 | 32 | 22
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 14 | 9 | 9
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 5 | 7
Headache (Nervous system disorders) | 16 | 16 | 18
Fatigue (General disorders) | 7 | 7 | 4
Pyrexia (General disorders) | 14 | 4 | 9
Folliculitis (Infections and infestations) | 5 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Rash papular (Skin and subcutaneous tissue disorders) | 3 | 5 | 1
Nausea (Gastrointestinal disorders) | 7 | 8 | 8
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 9
Vomiting (Gastrointestinal disorders) | 4 | 8 | 5
Dyspepsia (Gastrointestinal disorders) | 3 | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 9 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 9 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 10 | 8
Dizziness (Nervous system disorders) | 4 | 6 | 2
Asthenia (General disorders) | 3 | 5 | 2
Non-cardiac chest pain (General disorders) | 1 | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 7 | 4 | 6
Blood cholesterol increased (Investigations) | 5 | 4 | 5
Amylase increased (Investigations) | 5 | 3 | 1
Blood triglycerides increased (Investigations) | 5 | 1 | 2
Insomnia (Psychiatric disorders) | 5 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT02467270/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT02467270/SAP_001.pdf